CLINICAL TRIAL: NCT03872882
Title: Equipment Evaluation for Newborn Hearing Screening. A Randomised Comparison of Screen Outcome Between Standard Madsen 'Accuscreen New' and Madsen 'Accuscreen New' With Fast Refer Disabled and Increased Test Time
Brief Title: Accuscreen Equipment Evaluation For Newborn Hearing Screening
Status: Completed | Type: Observational
Sponsor: Julie Dawson (Other)
Collaborators: University of East Anglia (Other); GN Otometrics (Unknown)
Responsible Party: Sponsor-Investigator, Julie Dawson, Research Services Manager, Norfolk and Norwich University Hospitals NHS Foundation Trust
Organization: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Other Study IDs: 214416
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Hearing Loss
Keywords: Newborn hearing screening; Hearing loss; Hearing screening equipment
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An evaluation and comparison of results between the 'Accuscreen New' currently in use and an 'Accuscreen New' with different settings to see if the new settings reduce unnecessary referrals for babies from newborn hearing screening.

Babies will be tested with the standard and modified equipment. Referrals for diagnostic testing will be based on the standard equipment. A comparison in referrals between the standard and modified equipment will be made.

DETAILED DESCRIPTION:
All newborn babies undergo hearing screening, usually within the first few days of life and some are tested with the automated auditory brainstem response test (AABR). This involves recording activity from the hearing nerve and parts of the brainstem from three small sensors placed on the baby's head and neck when a series of clicking sounds are played in to the ear.

In March 2015 we started using an 'Accuscreen New' to record the AABR, which is approved by the Newborn Hearing Screening Programme (NHSP) and used widely across the UK. However, since introducing the new equipment the 'screen refer' rate increased significantly in very young babies (less than 48 hours old) and diagnostic testing showed they had satisfactory hearing. The impact of the increased referral rate caused increased delays on diagnostic testing and also lead to unnecessarily increased parental anxiety in relation to the hearing of their new born baby.

The equipment suppliers (GN Otometrics) and the NHSP Programme centre have agreed to an evaluation and comparison of results between the 'Accuscreen New' currently in use and an 'Accuscreen New' with different settings which we believe will reduce unnecessary referrals of so many young babies to Audiology (the modified equipment will test for up to 10 minutes to see if a response is present, instead of stopping after one or two minutes).

Babies will be tested with the standard and modified equipment. Referrals for diagnostic testing will be based on the standard equipment. A comparison in referrals between the standard and modified equipment will be made.

ELIGIBILITY:
Inclusion Criteria:

* Babies requiring AABR testing through newborn hearing screening

Exclusion Criteria:

-

Ages: 1 Day to 4 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Babies undergoing newborn hearing screening
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
Screen pass or screen refer | within 48 hours of birth
  The referral rate is the number of babies who do not pass the newborn hearing screen.

CONTACTS AND LOCATIONS:
Overall Officials: John Fitzgerald, BSc (Hons), Principal Investigator — Consultant Audiologist
Locations (1):
- Norfolk & Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No